CLINICAL TRIAL: NCT06203730
Title: Application of Dyadic Psychological Intervention Strategy Based on Double ABC-X Model in Patients With Maintenance Hemodialysis
Brief Title: Study on the Influence of Dyadic Psychoeducational Intervention on Patients With Maintenance Hemodialysis
Acronym: MHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Principal Investigator, Lijuan Zhou, Chief nurse, Jiangsu Taizhou People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYZhang
Record Dates: First submitted 2023-12-14; First posted 2024-01-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: double ABC-X model; MHD; quality of life; dyadic psychological intervention strategy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (No Intervention): The Blood purification Center provides routine care for MHD patients
- dyadic psychological intervention strategy (Experimental): an intervention strategy for both patients and caregivers that combines psychotherapy techniques and health management
  Interventions: Behavioral: dyadic psychological intervention strategy

INTERVENTIONS:
Behavioral: dyadic psychological intervention strategy — an intervention strategy for both patients and caregivers that combines psychotherapy techniques and health management
  Arms: dyadic psychological intervention strategy

SUMMARY:
This study aims explored the effectiveness of dual psychological intervention strategies in improving the quality of life of MHD patients based on the theoretical guidance of double ABC-X model. To provide a scientific and effective dual psychological intervention strategy for MHD patients and their caregivers, in order to improve the quality of life of MHD patients, and to provide a reference for nurses in clinical blood purification centers to implement psychological intervention.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of MHD patients were: (1) meeting the diagnostic criteria of CKD; (2) Maintenance hemodialysis at the blood purification center of our hospital for more than 3 months; (3) over 18 years of age; (4) Volunteer to participate in this study.
* MHD caregiver inclusion criteria: (1) over 18 years of age; (2) Responsible for the main care tasks of MHD patients; (3) Volunteer to participate in this study.

Exclusion Criteria:

* Exclusion criteria for MHD patients: (1) Patients with cognitive impairment or audio-visual impairment unable to communicate normally; (2) Patients diagnosed with mental illness or who are receiving medication or psychotherapy for depression.
* MHD caregiver exclusion criteria: (1) Caregivers with cognitive impairment or audiovisual impairment unable to communicate normally; (2) Caregivers suffering from serious heart, brain, liver, kidney and other important organ diseases; (3) carers or paid carers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
quality of life of patients with MHD | "Baseline" and "Immediately after the intervention"
  The Kidney Disease Quality of Life 36-item Short Form (KDQOL-36™) was used to measure quality of life in patients with MHD
anxiety of patients with MHD | "Baseline" and "Immediately after the intervention"
  The hospital anxiety and depression scale (HADS) was used to measure anxiety in patients with MHD
depression of patients with MHD | "Baseline" and "Immediately after the intervention"
  The hospital anxiety and depression scale (HADS) was used to measure depression in patients with MHD

SECONDARY OUTCOMES:
anxiety of caregivers burden | "Baseline" and "Immediately after the intervention"
  The hospital anxiety and depression scale (HADS) was used to measure anxiety in caregivers
depression of caregivers | "Baseline" and "Immediately after the intervention"
  The hospital anxiety and depression scale (HADS) was used to measure depression in caregivers
caregivers'burden | "Baseline" and "Immediately after the intervention"
  The Zarit Caregiver Burden Interview (ZBI) was used to measure caregivers' burden
Caregiving competence of caregivers | "Baseline" and "Immediately after the intervention"
  The Caregiving Competence Scale (CCS) was used to measure caregiving competence of caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou People's Hospital, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Zhang L, Chen Y, Tang W, Wang Q, Zou L, Zhou L. Effects of dyadic psychoeducational interventions for haemodialysis patients and their family caregivers: a randomised controlled trial. BMC Nurs. 2025 Mar 4;24(1):244. doi: 10.1186/s12912-025-02835-1. PMID 40038667